CLINICAL TRIAL: NCT02050841
Title: An Open-label, Multicenter, Post-Marketing Requirement (PMR) Study to Investigate the Safety, Tolerability and Efficacy of Octaplas in the Management of Pediatric Patients Who Require Replacement of Multiple Coagulation Factors.
Brief Title: Octaplas Pediatric Plasma Replacement Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAS-212
Record Dates: First submitted 2014-01-21; First posted 2014-01-31 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Liver Surgery; Liver Dysfunction; Coagulopathy; Cardiac Surgery
Keywords: Pediatric; patients; replacement; coagulation factors; plasma; s/d plasma; Octaplas; plasma replacement
MeSH Terms: conditions — Liver Diseases; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Octaplas (Experimental): Qualified patients will receive Octaplas as per protocol.
  Interventions: Biological: octaplas

INTERVENTIONS:
Biological: octaplas — Octaplas S/D Plasma

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and efficacy of octaplas in pediatric patients who require replacement of multiple coagulation factors. Replacement of multiple coagulation factors in pediatric patients with acquired deficiencies due to liver disease and/or in pediatric patients requiring cardiac surgery or liver surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring liver or cardiac surgery and/or patient with liver dysfunction associated with coagulopathy in whom replacement of multiple coagulation factors is required.
2. Voluntarily given, written and signed informed consent by the patient's legal representative(s) or guardian(s). Children deemed old enough by the Investigator/institution to understand the risks and benefits of the study should also be made aware of the risks/benefits of the study and provide written assent.
3. Male or female patient ≤ 16 years of age.

Exclusion Criteria:

1. Patient with known homozygous congenital deficiency of protein S.
2. Patient has a history of hypersensitivity reaction to blood or plasma-derived products or to any excipient of the investigational product.
3. Patient has an already known IgA (Immunoglobulin A) deficiency with documented antibodies against IgA.
4. Patient has a congenital factor deficiency or platelet disorder requiring plasma treatment.
5. Patient is currently participating in another study investigating a new drug product or another interventional clinical study that may impact coagulation factors or has participated during the last three (3) months.
6. Patient received FFP (Fresh Frozen Plasma), FP24 (Plasma frozen within 24 hours of collection) or any other plasma product other than Octaplas within the last 72 hours (cryoprecipitate and albumin are not exclusionary) prior to first Octaplas infusion.
7. Patient is on ECMO (Extracorporeal Membrane Oxygenation) when plasma is ordered by the treating physician for the first infusion episode.
8. Patient is pregnant.
9. Patient is predicted to require massive blood transfusion defined as more than 40 mL per kilogram of all blood products in a 24-hour period
10. Patient is receiving plasma exchange, therapeutic plasma exchange (TPE) or plasmapheresis.
11. Patient is a premature neonate defined as less than 37 weeks gestation.
12. Cardiac surgery patients who develop the need for plasma replacement greater than 72 hours after the end of the associated cardiac surgery and do not have coagulopathy due to hepatic dysfunction.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Study Director — International Medical Director
Locations (4):
- United States (4):
  - Octapharma Research Site, Birmingham, Alabama
  - Octapharma Research Site, Atlanta, Georgia
  - Octapharma Research Site, Minneapolis, Minnesota
  - Octapharma Research Site, St Louis, Missouri

REFERENCES:
- [Derived] Spinella PC, Borasino S, Alten J. Solvent/Detergent-Treated Plasma in the Management of Pediatric Patients Who Require Replacement of Multiple Coagulation Factors: An Open-Label, Multicenter, Post-marketing Study. Front Pediatr. 2020 Sep 17;8:572. doi: 10.3389/fped.2020.00572. eCollection 2020. PMID 33042916

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octaplas
Started | 50
Completed | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Octaplas
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.0 (3.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
ABO Blood Group [Count of Participants; unit: Participants]
  A | 16
  B | 9
  AB | 4
  O | 21
Height [Mean (Standard Deviation); unit: centimeters] | 78.1 (30.49)
Weight [Mean (Standard Deviation); unit: kilograms] | 13.66 (21.589)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 16.88 (5.421)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions (e.g., Allergic Reactions, TEs, TEEs (Thromboembolic Events) and Hyperfibrinolytic Events)
Time Frame: up to 6 days
Measure: Number; unit: participants
Arm/Group | Octaplas
Number analyzed (Participants) | 50
participants
  Any SAE | 5
  Any SAE related to Octaplas | 0
  Any ADR | 0
  Any ADR, SAE, HFE TEE, or TE leading to withdrawal | 0
  Any ADR, SAE, HFE, TEE, or TE leading to death | 1
  Any study death related to Octaplas | 0

2. Primary Outcome: Monitoring of Clinically Significant Changes in White Blood Cells
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: 10^3/µL
Groups:
- Children >2 Years; Infants ≤2 Years: Qualified patients will receive Octaplas as per protocol.
  octaplas: Octaplas S/D Plasma
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
10^3/µL | 5.3 [-4.7 to 28.3] | 2.05 [-12.3 to 9.3]

3. Primary Outcome: Monitoring of Clinically Significant Changes in Red Blood Cells
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: 10^6/µL
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
10^6/µL | -0.34 [-1.4 to 0.6] | -0.06 [-1.8 to 1.8]

4. Primary Outcome: Monitoring of Clinically Significant Changes in Hemoglobin
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: g/dL
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
g/dL | -0.70 [-3.9 to 2.7] | 0.80 [-4.6 to 5.2]

5. Primary Outcome: Monitoring of Clinically Significant Changes in Hematocrit
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: volume percentage of RBC in blood
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
volume percentage of RBC in blood | -2.35 [-10.8 to 6.5] | 1.35 [-14.6 to 16.2]

6. Primary Outcome: Monitoring of Clinically Significant Changes in Mean Corpuscular Volume (MCV)
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: fL
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
fL | 1.6 [-5.4 to 6.3] | 1.85 [-22.8 to 9.1]

7. Primary Outcome: Monitoring of Clinically Significant Changes in Mean Corpuscular Hemoglobin (MCH)
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: pg
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
pg | 0.85 [-1.8 to 2.9] | 1.00 [-8.3 to 5.6]

8. Primary Outcome: Monitoring of Clinically Significant Changes in Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: g/dL
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
g/dL | -0.15 [-0.9 to 4.2] | 0.20 [-1.2 to 2.8]

9. Primary Outcome: Monitoring of Clinically Significant Changes in Red Cell Distribution Width (RDW)
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: % variation of RBC size
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
% variation of RBC size | 0.10 [-3.9 to 3.0] | 0.40 [-2.1 to 4.2]

10. Primary Outcome: Monitoring of Clinically Significant Changes in Platelets
Description: Assesses Pre- and Post-infusion for Infusion Episode 1
Time Frame: up to 6 days
Measure: Median (Full Range); unit: 10^3/µL
Arm/Group | Children >2 Years | Infants ≤2 Years
Number analyzed (Participants) | 13 | 37
10^3/µL | -105.5 [-210.0 to 15.0] | -167.00 [-410.0 to 215.0]

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hemostatic Parameters as Measured by the Following: International Normalized Ratio (INR)
Description: This hemostatic parameter is figured out in the lab and helps to diagnose a bleeding disorder or excessive clotting disorder. The change of INR before and after 1st Octaplas infusion was scrutinized by analyzing the shifts between the classifications given below.
Time Frame: up to 6 days
Measure: Number; unit: participants
Arm/Group | Octaplas
Number analyzed (Participants) | 50
participants
  Shift from Not Clinically Significant to Normal | 1
  Remained Normal | 8
  Remained Not Clinically Significant | 11
  Shift from Normal to Not Clinically Significant | 25
  Shift to or from Clinically Significant | 1

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hemostatic Parameters as Measured by the Following: Prothrombin Time (PT)
Description: This hemostatic parameter is figured out in the lab and measures the time it takes for your blood to clot (the higher the PT the longer it takes your blood to clot). The change of PT before and after 1st Octaplas infusion was scrutinized by analyzing the shifts between the classifications given below.
Time Frame: up to 6 days
Measure: Number; unit: participants
Arm/Group | Octaplas
Number analyzed (Participants) | 50
participants
  Shift from Not Clinically Significant to Normal | 1
  Remained Normal | 8
  Remained Not Clinically Significant | 18
  Shift from Normal to Not Clinically Significant | 19
  Shift to or from Clinically Significant | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hemostatic Parameters as Measured by the Following: Thromboelastography (TEG) or Thromboelastometry (ROTEM).
Description: TEG and ROTEM are methods of testing the efficiency of blood coagulation. The results were compared by looking at potential trends from TEG and ROTEM between pre-infusion vs post-infusion time points.
Time Frame: up to 6 days
Measure: Number; unit: participants
Groups:
- EPL30-TEG: Number of Participants With Clinically Significant Changes in Hemostatic Parameters as Measured by EPL30-TEG (estimated percent lysis)
- ML30-ROTEM: Number of Participants WithClinically Significant Changes in Hemostatic Parameters as Measured byThromboelastometry (ROTEM).
Arm/Group | EPL30-TEG | ML30-ROTEM
Number analyzed (Participants) | 50 | 50
participants
  Shift from Not Clinically Significant to Normal | 1 | 0
  Remained Normal | 40 | 0
  Remained Not Clinically Significant | 0 | 0
  Shift from Normal to Not Clinically Significant | 0 | 0
  Shift to or from Clinically Significant | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hemostatic Parameters as Measured by the Following: Activated Partial Thromboplastin Time (aPTT)
Description: aPTT measures the length of time (in seconds) that it takes for clotting to occur in a test cube. The higher the number of seconds the longer it takes the blood to clot. The changes between pre - and post infusion were analyzed
Time Frame: up to 6 days
Measure: Number; unit: participants
Arm/Group | Octaplas
Number analyzed (Participants) | 50
participants
  From (NCS) Not Clinically Significant to Normal | 5
  Remained Normal | 18
  Remained Not Clinically Significant (NCS) | 12
  Shift from Normal to Not Clinically Significant | 9
  NCS to Clinically Significant Shift | 1
  Clinically Significant to NCS shift | 1

15. Secondary Outcome: Volume (Dose in mL/kg) of Octaplas Used Per Infusion Episode for Each Patient.
Description: Normal infusion: Replacement of multiple clotting factors Bypass priming: Limit hemodilution and reduce transfusion requirements Bypass warming up: Rewarm patients suffering from hypothermia during the surgery process
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Octaplas
Number analyzed (Participants) | 50
mL/kg
  Normal Infusion | 15 (14.17)
  Bypass Priming | 20.2 (7.82)
  Bypass Warming Up | 15.9 (5.88)

16. Secondary Outcome: Medically Significant Changes in Blood Pressure
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: mm of Hg
Groups:
- Octaplas - Pre-Infusion: Pre-Infusion Vital Signs
- Octaplas - Post-Infusion: Post-Infusion Vital Signs
Arm/Group | Octaplas - Pre-Infusion | Octaplas - Post-Infusion
Number analyzed (Participants) | 50 | 50
mm of Hg
  Systolic Blood Pressure | 75.66 (16.901) | 79.96 (16.437)
  Diastolic Blood Pressure | 46.28 (10.031) | 50.00 (11.648)

17. Secondary Outcome: Medically Significant Changes in Heart Rate
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Octaplas - Pre-Infusion | Octaplas - Post-Infusion
Number analyzed (Participants) | 50 | 50
beats per minute | 122.86 (30.528) | 132.80 (24.439)

18. Secondary Outcome: Medically Significant Changes in Respiratory Rate
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Octaplas - Pre-Infusion | Octaplas - Post-Infusion
Number analyzed (Participants) | 50 | 50
breaths/minute | 21.27 (7.335) | 23.79 (6.702)

19. Secondary Outcome: Medically Significant Changes in Oxygen Saturation
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: % oxygen in blood
Arm/Group | Octaplas - Pre-Infusion | Octaplas - Post-Infusion
Number analyzed (Participants) | 50 | 50
% oxygen in blood | 96.86 (5.564) | 98.33 (3.204)

20. Secondary Outcome: Medically Significant Changes in Body Temperature
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Octaplas - Pre-Infusion | Octaplas - Post-Infusion
Number analyzed (Participants) | 50 | 50
units | 35.60 (2.023) | 36.50 (1.597)

21. Secondary Outcome: Count of Investigator's Assessment of Overall Safety Observed for Patients by Category (Assessed to Have Overall Safety of 'Excellent', Assessed to Have Overall Safety of 'Moderate', Assessed to Have Overall Safety of 'Poor')
Time Frame: up to 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplas
Number analyzed (Participants) | 50
Participants
  Assessed to have overall safety of 'excellent' | 50
  Assessed to have overall safety of 'moderate' | 0
  Assessed to have overall safety of 'poor' | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant over the course of 6 days
Description: Any of the following drug safety information was collected after the start of the first infusion episode:
  * Serious adverse events
  * Adverse drug reactions temporally associated with administration of the investigational product
  * Adverse events that fall into the category of TEs, TEEs and hyperfibrinolytic events
  * Post-treatment related safety reports, pregnancies, drug overdose, interaction, abuse, misuse, medication error, lack of efficacy
Arm/Group | Octaplas
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 5/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplas (N=50)
Portal vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Iatrogenic injury (Surgical and medical procedures) | 1 (1)
Haemorrhage coronary artery (Vascular disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT02050841/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT02050841/SAP_001.pdf